CLINICAL TRIAL: NCT02450110
Title: A Pilot Study of Spinal Cord Stimulation in Heart Failure Patients With Depressed Left Ventricular Function
Acronym: RAPID-HELP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unexpectedly slow recruitment rate
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAPID-HELP
Record Dates: First submitted 2015-05-12; First posted 2015-05-21 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Heart Failure; Systolic Dysfunction
Keywords: spinal cord stimulation; heart failure; autonomic regulation; BNP; left ventricle systolic dysfunction
MeSH Terms: conditions — Heart Failure | interventions — Spinal Cord Stimulation

ARMS (2):
- Intervention (Experimental): Spinal cord stimulation on top of standard treatment
  Interventions: Device: Spinal cord stimulation
- Control (No Intervention): Standard treatment

INTERVENTIONS:
Device: Spinal cord stimulation
  Arms: Intervention

SUMMARY:
A randomized pilot study of spinal cord stimulation in patients with chronic heart failure aiming to show whether this therapy impacts central haemodynamic and autonomic regulations.

DETAILED DESCRIPTION:
Patients will be randomized (1:1) for spinal cord stimulation as an addition to optimal guidelines-driven management or to control group on optimal management only. Spinal cord stimulation will be performed for 30 days, and outcome measures will be testes before stimulation, after 30 days stimulation and after 30 days of further follow-up. The control group will be studied at baseline and after 30 days only.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic heart failure II-III class (NYHA);
2. Age 18-70 years;
3. Left ventricle ejection fraction ≤35%;
4. Optimal heart failure management according to the guidelines;
5. Signed informed consent

Exclusion Criteria:

1. Heart transplant list;
2. Acute conditions, including systemic infection;
3. Reversible cause of heart failure (thyroid gland diseases, alcoholic intoxication etc);
4. Planned elective heart surgery or intervention;
5. Recent (3 months) myocardial infarction, coronary intervention;
6. Heart failure decompensation;
7. Implanted cardiac resynchronization device < 6 months ago;
8. Contraindications for lumbal puncture or placement of a spinal cord pacing electrode;
9. Permanent atrial fibrillation;
10. Stroke or TIA < 6 months ago;
11. Pulmonary thromboembolist < 3 months ago;
12. Hypertrophic cardiomyopathy with obstruction;
13. Angina III-IV class, or congestive heart failure IV class;
14. Participation in any other clinical trial;
15. Women of childbearing possibility without appropriate contraception, pregnant, or breastfeeding women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-02; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Dynamics of NT-pro-BNP-level | Baseline, 30, 60 days
  NT-pro-BNP-level baseline, 30 days and 60 days (intervention) NT-pro-BNP-level baseline, 30 days (control)

SECONDARY OUTCOMES:
Exercise capacity as determined by a cardiopulmonary test | Baseline, 30, 60 days
  Exercise capacity (cardiopulmonary test) baseline, 30 days and 60 days (intervention) Exercise capacity (cardiopulmonary test) baseline, 30 days (control)
Changes in heart failure functional class | Baseline, 30, 60 days
Changes in atrial effective refractory period | Baseline, 30, 60 days
Number of participants with ventricular arrhythmias | Baseline, 30, 60 days
Autonomic regulation tests results change | Baseline, 30, 60 days
  Tilt-test, Valsalva maneuver, deep breath test
Levels of pro-inflammatory plasma markers | Baseline, 30, 60 days
  TNF-a, CRP, fibrinogen
Changes in left ventricle ejection fraction as determined by echocardiography | Baseline, 30, 60 days
Left ventricle volume | Baseline, 30, 60 days
Number of participants with complications | Baseline, 30, 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny V Shlyakhto, MD, DSc, Principal Investigator — Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health
Locations (1):
- Federal North-West Medical Research Centre, Saint Petersburg, Russia